CLINICAL TRIAL: NCT05242133
Title: Efficacy and Safety of Peginterferon Beta-1a (CinnaGen) Versus CinnoVex® (CinnaGen) in Reducing the Annualized Relapse Rate in Participants With Relapsing Remitting Multiple Sclerosis: A Phase III, Randomized, Parallel, Noninferiority Study
Brief Title: Efficacy and Safety of Peginterferon Beta-1a (CinnaGen) in Participants With Relapsing Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cinnagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEG.CIN.AZ.94.III; IRCT201612306135N8 (Other: Food And Drug Administration of The Islamic Republic of Iran)
Record Dates: First submitted 2022-01-17; First posted 2022-02-16 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Relapsing Remitting Multiple Sclerosis (RRMS)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CinnaGen peginterferon beta-1a (Experimental): Pegylated interferon beta-1a (CinnaGen) autoinjector (Physioject™),125 mcg, subcutaneous (SC) injection, every 2 weeks, for 24 months
  Interventions: Drug: Pegylated interferon beta-1a
- CinnoVex® (Active Comparator): Interferon Beta-1A Prefilled Syringe, CinnoVex® (CinnaGen), 30 mcg, intramuscular injection, once a week, for 24 months
  Interventions: Drug: Interferon Beta-1A Prefilled Syringe

INTERVENTIONS:
Drug: Pegylated interferon beta-1a — Pegylated interferon beta-1a (CinnaGen) autoinjector (Physioject™),125 mcg, subcutaneous (SC) injection, every 2 weeks, for 24 months
  Arms: CinnaGen peginterferon beta-1a
Drug: Interferon Beta-1A Prefilled Syringe — Interferon Beta-1A Prefilled Syringe, CinnoVex® (CinnaGen), 30 mcg, intramuscular injection, once a week, for 24 months
  Other Names: CinnoVex®
  Arms: CinnoVex®

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of peginterferon beta-1a produced by CinnaGen compared with CinnoVex® (CinnaGen) in subjects with relapsing remitting multiple sclerosis (RRMS). All the participants will receive one of the following regimens: pegylated interferon beta-1a (CinnaGen), autoinjector (Physioject™), 125mcg, subcutaneous, every 2 weeks for 24 months or CinnoVex® (CinnaGen), prefilled syringes, 30mcg, intramuscular, once a week for 24 months. The primary objective of this study is to verify the non-inferiority of peginterferon beta-1a (CinnaGen) versus CinnoVex® (CinnaGen) in reducing the annualized relapse rate (ARR) in participants with relapsing remitting multiple sclerosis (RRMS) at 2 years.

The secondary objectives of this study are:

* Reducing the total number of new or newly enlarging T2 hyperintense lesions on brain magnetic resonance imaging (MRI) scans
* Slowing the progression of disability
* Comparing adverse events

DETAILED DESCRIPTION:
The purpose of this phase III, randomized, active control, parallel, non-inferiority, multicenter study is to verify the non-inferiority of peginterferon beta-1a produced by CinnaGen versus CinnoVex® (CinnaGen) in subjects with relapsing remitting multiple sclerosis (RRMS).

All the participants will receive one of the following regimens:

I. Pegylated interferon beta-1a (CinnaGen), autoinjector (Physioject™), 125mcg, subcutaneous, every 2 weeks for 24 months; II. Interferon beta-1a, CinnoVex® (CinnaGen), prefilled syringes, 30mcg, intramuscular, once a week for 24 months.

With the aim of ensuring the compliance and safety, in the first two months of the study, in each monthly visit, a trained expert nurse will be responsible for drug injection for both intervention groups and will train all patients for self-injection. By the end of the first two months to the end of the study, patients will self-inject the medication in both groups.

All other cares or medications will be allowed to continue by patients, except for disease modifying therapies (DMTs) and medicines which affect the immune system (e.g. immunosuppressants and immunomodulators). Any concomitant medication will be recorded for patients in their regular visits.

The primary objective of this study is to verify the non-inferiority of peginterferon beta-1a (CinnaGen) versus CinnoVex® (CinnaGen) in reducing the annualized relapse rate (ARR) in participants with relapsing remitting multiple sclerosis (RRMS) at 2 years.

The secondary objectives of this study are:

* Reducing the total number of new or newly enlarging T2 hyperintense lesions on brain magnetic resonance imaging (MRI) scans
* Slowing the progression of disability
* Comparing safety issues

Sample size:

Group sample sizes of 76 in the experimental group and 76 in the active comparator group will achieve almost 80% power to detect non-inferiority using a one-sided, two-sample t-test. The margin of non-inferiority is 0.17. The true ratio of the means at which the power is evaluated is 1.00. The significance level of the test is 0.05. The coefficients of variation of both groups are assumed to be 0.4. The dropout rate is assumed to be 10%; hence 168 patients will be randomized.

Sequence generation:

The randomization plan of the patients will be carried out centrally using Cran-R version 3.2.3. Using permuted block randomization, blocks (length of each block is 4 or 2) will be made, for a total of 168 patients with 1:1 allocation ratio. Once the randomization has been made, each patient is given a code with which he/she will be identified throughout the study. The assigned code will be made up of 3 numbers (corresponding to the randomization number) and by 4 initials (corresponding to the 2 first letter of the first name, the 2 first letter of the first surname) and 2 numbers (center code). The randomization number will be assigned in a consecutive way.

Blinding:

Because of the different routes of administration of drugs in the study groups, patient blinding is not possible.

Data management:

Principal investigator is responsible for safe keeping of all patients' records at all times. Original hard copies of case report forms (CRFs) will be sent to Clinical Trial Consultants (CTCs) upon request and at the end of the study for data management. A copy of the records will be kept at the center. Sending and receiving of all patients' documents will be made after taking into consideration safety and security issues.

Principal investigator should set necessary schemes to control the quality of:

* Drug delivery, storage and handling
* All clinical examinations
* Laboratory tests and other paraclinical investigations
* Patient care

Data monitoring:

The objectives of the data quality control (QC) are:

* To ensure the existence of the patients and the respect of ethics, including signed patient informed consent forms (ICFs)
* To identify the issues, including systematic issues, as early as possible for appropriate setting of action plans and corrective actions
* To ensure the validity of the data To meet these objectives, the possibility of the sites' QC must be explained to the investigators at the time of the study initiation and agreed by them. QC will be performed on sites by the Local Study Teams.

QC will be started after inclusion of 30% of patients and will be ended before 80% of inclusion.

Two levels of QC will be performed:

Quality of CRF completion: At the time of CRF reception, the Local Study Team will review the completed CRFs in order to assess the completeness and the quality of completion. The Local Study Team (monitor or designee) is responsible to set up an action plan in order to improve the quality at site level. In case of systematic issue, the Local Study Team will inform the Corporate Study Team.

Central database checks: In addition to the standard data management activities, the following parameters will be systematically assessed as a part of the QC of the study, in country- and site-levels by the Study Central Team:

* Signed ICFs
* Rates of error and missing data for the key variables
* Completion of the patients' questionnaire
* Enough clarity of the forms During the QC visit, the monitor will have to complete a QC visit report.

Principal investigators should set necessary schemes to control the quality of:

* Signed ICF
* Drug delivery, storage and handling
* All clinical examinations
* Laboratory tests and other paraclinical investigations
* Patient care

Research ethics approval:

* Ethics committee approval is mandatory for this study to commence.
* No patient will be recruited to this study without an informed consent.
* It will be made clear to all patients that they can leave the study any time they desire with no need for any explanation.
* To keep confidentiality in case of a lost document, the name and surname of the patients will not appear on evaluation forms.
* Adverse effect report forms will be processed after each visit. Research team is responsible for dealing with immediate aftermath of any adverse event regardless of whether or not the event is directly related to the medication that is being studied.
* All serious adverse events should be reported to DSMB (Data and Safety Monitoring Board). The board is responsible for making necessary decisions to deal with the situation. These decisions may include determining the relationship between the drug and the observed adverse event.
* The protocol, CRF, information for patients and informed consent forms will be submitted to the ethics committees responsible for the investigators in TUMS, for review and approval according to the national regulatory guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting multiple sclerosis diagnosis (based on McDonald criteria 2010)
* Expanded Disability Status Scale between 0 to 5
* At least one relapse having occurred within the past 12 months.
* Subjects have refused alternative treatments and other available therapies
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent
* Negative pregnancy test for women of childbearing age

Exclusion Criteria:

* Primary progressive, secondary progressive, or progressive relapsing MS
* Female subjects considering becoming pregnant while in the study or currently breastfeeding
* Subjects for whom MRI was contraindicated, i.e., who had pacemakers or other contraindicated implanted metal devices, were allergic to gadolinium, or had claustrophobia that could not be medically managed.
* Unwillingness or inability to comply with the requirements of the protocol including the presence of any condition (physical, mental or social) that was likely to affect the subject's ability to comply with the protocol.
* Pre-speciﬁed laboratory abnormalities
* History of any clinically significant (as determined by the Investigator) cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal, or other major disease that would preclude participation in a clinical trial.
* History of malignant disease, including solid tumors and hematologic malignancies (with the exception of basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured).
* History of seizure disorder or unexplained blackouts or history of a seizure within 3 months prior to baseline.
* History of suicidal ideation within 3 months prior to Baseline or an episode of severe depression within 3 months prior to Baseline. Severe depression is defined as an episode of depression that requires hospitalization, or at the discretion of the Investigator.
* Abnormal screening blood tests exceeding any of the limits defined below:

  * Alanine transaminase/serum glutamate pyruvate transaminase (ALT/SGPT) greater than 2 times the upper limit of normal (>2 × ULN) or aspartate transaminase/serum glutamic oxaloacetic transaminase (AST/SGOT) >2 × ULN or bilirubin >1.5 × ULN.
  * Total white blood cell count (WBC) <4000 /mm3
  * Absolute Neutrophil Count (ANC) of < 1500 /mm3
  * Platelet count <150,000 c/mm3
  * Hemoglobin <10 g/dL in female subjects; <11 g/dL in male subjects
  * Serum creatinine> upper limit of normal lab value
* A MS relapse that has occurred within the 30 days prior to randomization and/or the subject has not been stabilized from a previous relapse prior to randomization (Day 1).
* Elective surgery performed within 2 weeks prior to randomization (Day 1) or scheduled to be performed through the study interval.
* Treatment with other agents to treat MS symptoms or underlying disease as specified below:
* Agent Time Required off Agent Prior to Baseline:

  * Any prior treatment with:

    * Total Lymphoid Irradiation
    * Cladribine
    * T-cell Vaccine
    * Natalizumab
    * Rituximab
    * Plegridy®
  * Prior treatment within 1 year of randomization:

    * Cyclophosphamide
    * Mitoxantrone
  * Prior treatment within 6 months prior to randomization:

    * Cyclosporine
    * Plasma exchange
    * Intravenous immunoglobulin (IVIG)
    * Azathioprine
    * Methotrexate
  * Subjects must have discontinued interferon treatment at least 6 months prior to randomization
  * Prior treatment within 30 days prior to randomization:

    - Systemic corticosteroids
  * Prior treatment with glatiramer acetate within 4 weeks prior to randomization
  * Treatment with another investigational drug or approved therapy for investigational use within the 6 months prior to randomization
  * Other unspecified reasons that, in the opinion of the Investigator, made the subject unsuitable for enrolment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Annualized Relapse Rate | 96 weeks
  The total number of relapses divided by the total person-time at risk of relapse. A relapse is defined as the appearance of a new or worsening of a previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding relapse. The abnormality must be present for at least 24 hours and occur in the absence of fever or infection.

SECONDARY OUTCOMES:
Proportion of patients with 12 weeks of sustained disability progression | Baseline up to week 96
  Clinical evaluation
Total number of new or newly enlarging T2-hyperintense lesions as detected by brain MRI | Baseline up to week 96
  Sum of the individual number of new or newly enlarging T2-hyperintense lesions at weeks 24, 48, and 96
Total number of gadolinium enhancing lesions as detected by brain MRI | Baseline up to week 96
  Sum of the individual number of gadolinium enhancing lesions at weeks 24, 48, and 96
Total number of new or newly enlarging T1 hypointense lesions as detected by brain MRI | Baseline up to week 96
  Sum of the individual number new T1 hypointense lesions at weeks 24, 48, and 96
Total number of new active lesions as detected by brain MRI | Baseline up to week 96
  Sum of gadolinium enhancing plus non-enhancing new or newly enlarging T2 hyperintense lesions
Volume of new or newly enlarging T2 hyperintense lesions as detected by brain MRI | Baseline up to week 96
  Inflammatory activity based on MRI measurement of new or newly enlarging T2 lesion volume
Volume of gadolinium enhancing lesions as detected by brain MRI | Baseline up to week 96
  Inflammatory activity based on MRI measurement of gadolinium enhancing T1 lesion volume
Volume of new or newly enlarging T1 hypointense lesions as detected by brain MRI | Baseline up to week 96
  Inflammatory activity based on MRI measurement of hypointense T1 lesion volume
Brain atrophy | Baseline up to week 96
  Percentage of brain volume change from baseline detected by brain MRI

OTHER OUTCOMES:
Number of participants with Adverse Events (AEs) | 96 weeks
  Intensity, seriousness and causality assessment of observed AEs, and abnormal laboratory findings

CONTACTS AND LOCATIONS:
Locations (1):
- Sina Hospital, Tehran, Iran

REFERENCES:
- [Background] Calabresi PA, Kieseier BC, Arnold DL, Balcer LJ, Boyko A, Pelletier J, Liu S, Zhu Y, Seddighzadeh A, Hung S, Deykin A; ADVANCE Study Investigators. Pegylated interferon beta-1a for relapsing-remitting multiple sclerosis (ADVANCE): a randomised, phase 3, double-blind study. Lancet Neurol. 2014 Jul;13(7):657-65. doi: 10.1016/S1474-4422(14)70068-7. Epub 2014 Apr 30. PMID 24794721
- [Background] National Multiple Sclerosis Society. (2017). FDA Approves Plegridy (Pegylated Interferon Beta) For Relapsing MS. [online] Available at: http://www.nationalmssociety.org/About-the-Society/News/FDA-Approves-Plegridy-Pegylated-Interferon-Beta [Accessed 2 Sep. 2017].
- [Background] Anon, (2017). [online] Available at: http://www.cinnagen.com/index.php/our-products/human-medicines/cinnovex [Accessed 2 Sep. 2017].
- [Background] Anon, (2017). [online] Available at: National Multiple Sclerosis Society. (2017). FDA Approves Plegridy (Pegylated Interferon Beta) For Relapsing MS. [online] Available at: http://www.nationalmssociety.org/About-the-Society/News/FDA-Approves-Plegridy-Pegylated-Interferon-Beta. [Accessed 2 Sep. 2017].
- [Derived] Shaygannejad V, Ashtari F, Saeidi M, Beladi Moghadam N, Ghalyanchi Langroodi H, Baghbanian SM, Abolfazli R, Ghiasian M, Ayromlou H, Asadollahzadeh E, Sabzvari A, Kafi H, Azimi Saeen A. Efficacy and safety of peginterferon beta-1a compared to interferon beta-1a in relapsing remitting multiple sclerosis patients: A phase 3, randomized, non-inferiority clinical trial (PEGINTEGRITY). Mult Scler Relat Disord. 2024 Oct;90:105839. doi: 10.1016/j.msard.2024.105839. Epub 2024 Aug 20. PMID 39217809